CLINICAL TRIAL: NCT07176455
Title: Research on the Temporal Transformation Mechanism and Intervention Strategies of Frail-related Dietary Behaviors in Older Gastric Cancer Survivors
Brief Title: Temporal Transformation Mechanism and Intervention Strategies of Frail-related Dietary Behaviors in Older Gastric Cancer Survivors
Status: Enrolling by invitation | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yinning Guo, Principal Investigator, Nanjing Medical University
Other Study IDs: 2025-79
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Gastric Cancer (GC); Frailty in Adult Surgery
Keywords: gastric cancer; frailty; dietary behavior
MeSH Terms: conditions — Stomach Neoplasms; Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Frail-promoting dietary behavior group
  Interventions: Behavioral: Anti-frailty dietary behavior intervention

INTERVENTIONS:
Behavioral: Anti-frailty dietary behavior intervention — Design intervention measures based on the mechanism of dietary behavior changes related to frailty

SUMMARY:
The investigators invite participants to participate in the research project "Research on the Maintenance Mechanism and Intervention Strategies of Dietary Behavior Changes Related to Frailty in Elderly Gastric Cancer Survivors". This project is funded by the School of Nursing of Nanjing Medical University and will be carried out in the Gastroenterology Department of the General Surgery Department of the First Affiliated Hospital of Nanjing Medical University and the Affiliated Cancer Hospital of Nanjing Medical University. Participants have been invited to join this research because participants meet the inclusion criteria for the study.

This informed consent form provides participants with some information to help participants decide whether to participate in this clinical study. Participants' participation in this study is voluntary. This research has been reviewed and approved by the Ethics Committee of Nanjing Medical University. If participants agree to join this study, please refer to the following instructions. Please read carefully. If participants have any questions, please raise them to the researcher in charge of this study.

Research objective (Why conduct this research?) China is a country with a high incidence of gastric cancer. Its incidence and mortality rates both rank among the top five in the world, seriously endangering the health of its citizens. With the intensification of aging, the proportion of gastric cancer patients over 60 years old among all gastric cancer patients has reached as high as 75.2%, making elderly gastric cancer patients a large group. Nutrition plays a crucial role in the frailty development of elderly survivors of gastric cancer.

Research process and methods (What needs to be done if participating in the research?) If participants are willing to participate in this study, participants will be surveyed at the time points of discharge and 1 month, 3 months and 6 months after the operation. During participants' hospitalization (at admission and discharge), the investigators will use the Sociodemographic and Physiological Pathological Questionnaire, the Dietary Behavior Scale, the Tilburg Frailty Scale, the Depression-Anxiety-Stress Scale, the Family Nutrition Behavior Health Action Process Scale for Postoperative Gastric Cancer Patients, the Family Care Index Evaluation Scale, the Perceived Social Support Scale, the Family Food Environment Scale, and the Policy Environment Questionnaire to investigate participants Relevant variable indicators; At 1 month, 3 months and 6 months after the operation, telephone follow-up will be conducted using the Eating Behavior Scale, Tilburg Frailty Scale, Depression-anxiety-Stress Scale, Family Nutrition Behavior Health Action Process Scale for Postoperative Gastric Cancer Patients, Family Care Index Rating Scale, Perceived Social Support Scale and Family Food Environment Scale to dynamically evaluate the scores of relevant variables. It is used for the extraction of dietary behaviors related to later frailty and the exploration of the maintenance mechanism of transformation.

What are the possible benefits of participating in the research? During the longitudinal telephone follow-up, the investigators can answer some of your questions and provide health assistance to participants. Meanwhile, the research results of this study are beneficial for later dietary nutrition and frailty management.

What are the possible risks of participating in the research? The above-mentioned survey poses no risk to participants' health or prognosis recovery.

Do participants need to pay any relevant fees to participate in the research? There is no need to pay any related fees to participate in this study.

Is personal privacy kept confidential? The data in this study may be published, but participants' personal privacy-related information will be strictly confidential.

Must participants take part in the research? Participation in this research is completely voluntary. Participants can refuse to take part in the research or withdraw from it at any stage of the research process. The investigators sincerely hope that participants will contribute to scientific research. However, whether participants participate or not, the investigators will respect participants' choice and guarantee that it will not have any impact on participants' diagnosis, treatment and care. If participants decide to participate in this study, please sign this informed consent form.

If participants have any questions related to participants' personal rights and interests, participants can contact the Ethics Committee of Nanjing Medical University. The contact number is 025-86869212.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gastric cancer; Performed the radical gastrectomy; Discharge within one month after surgery; Age ≥60 years old; Aware of personal diagnosis; Must be able to articulate views clearly; Voluntarily agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

* Severe cardiac, hepatic, pulmonary, or renal insufficiency; Tumors in other sites.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing radical gastrectomy for gastric cancer at selected tertiary hospitals in Jiangsu Province between July 2025 and October 2026 were enrolled as study subjects. Discharge served as the baseline (T0), with follow-up surveys conducted at 1 month post-surgery (T1), 3 months post-surgery (T2), and 6 months post-surgery (T3).
Sampling Method: Probability Sample
Enrollment: 438 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
frailty:frailty was measured using the Tilburg frailty indicator (TFI). It consists of 15 items across three domains, scores range from 0 to 15, with higher scores indicating greater frailty; a score ≥5 denotes frailty. | The first month, the third month and the sixth month after radical gastrectomy for gastric cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No
This was applied for by all of us together. Everyone is clear about the research plan, so there is no need to share the IPD again